CLINICAL TRIAL: NCT00579254
Title: Real Life Experience With Caduet Evaluating Effectiveness, Safety and Tolerability in the Management of Cardiovascular Risk Factors (EXCEL Study)
Brief Title: Real Life Experience With Caduet In Patients With Cardiovascular Risk Factors
Acronym: EXCEL
Status: Terminated | Type: Observational
Why Stopped: See the termination reason in detailed description.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A3841054
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Results first posted 2009-06-19 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Hypertension and Cardiovascular Risk Factors
Keywords: Efficacy,safety & tolerability of Caduet In Patients With Cardiovascular Risk Factors
MeSH Terms: conditions — Hypertension | interventions — amlodipine, atorvastatin drug combination; Amlodipine; Atorvastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CADUET (AMLODIPINE 5 mg/ATORVASTATIN 10 mg or 20 mg) — Patients who have been treated with Caduet 5/10 or 5/20 mg single pill treatment, based on their clinical conditions and latest locally approved packet insert recommendations will be eligible to be enrolled to this study

SUMMARY:
To assess the effect of single pill therapy on the management of hypertension and other cardiovascular risk factors (e.g., dyslipidemia) in Indian patients in whom the treating doctor has already considered that the administration of the amlodipine/atorvastatin single pill to be appropriate

DETAILED DESCRIPTION:
Patients who have been prescribed single pill Caduet are eligible to participate in this study. The treating physician will obtain written informed consent from each subject or the subject's legally acceptable representative before any study-specific activity is performed.

The study terminated on May 5, 2008. The decision to terminate was due to inability to achieve study timelines and undue delay in obtaining IEC/IRB permission at some sites. No safety or efficacy issues caused the decision to terminate.

ELIGIBILITY:
Inclusion Criteria:

Patients who have been prescribed single pill Caduet are eligible to participate in this study. Patients will be treated in this study according to prevailing local clinical practice following the locally approved product labeled recommendations.

Exclusion Criteria:

* Known hypersensitivity to dihydropyridines, amlodipine, atorvastatin, or any component of this medication,
* Active liver disease or unexplained persistent elevations of serum transaminases exceeding three times the upper limit of normal,
* Or who are pregnant, breast-feeding, or of childbearing potential who are not using adequate contraceptive measures. Amlodipine/atorvastatin should be administered to women of childbearing age only when such patients are highly unlikely to conceive and have been informed of the potential hazards to the fetus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be treated in this study according to prevailing local clinical practice following the locally approved product labeled recommendations
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2007-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3841054&StudyName=Real%20Life%20Experience%20With%20Caduet%20In%20Patients%20With%20Cardiovascular%20Risk%20Factors

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a phase 4, observational, open-label study conducted in patients who were prescribed singlepill Caduet by their treating physician per usual clinical practice. Study drug was not provided by the Sponsor.
Groups:
- Caduet: Patients were treated with Caduet (5/10 or 5/20 mg) in this study according to prevailing local clinical practice following the locally approved product labeled recommendations.
Period: Overall Study
Arm/Group | Caduet
Started | 112
Completed | 0
Not Completed | 112
Not completed — Lost to Follow-up | 39
Not completed — Discontinued when study terminated | 73

BASELINE CHARACTERISTICS:
Arm/Group | Caduet
Number analyzed (Participants) | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 71

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic and Diastolic Blood Pressure
Description: No efficacy results were available from this terminated study.
Time Frame: Baseline, 24 weeks
Arm/Group | Caduet
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Caduet
Serious Adverse Events (participants affected / at risk) | 0/112
Other Adverse Events (participants affected / at risk) | 1
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Caduet
High Density Lipoprotein decreased (Investigations) | 1/112

LIMITATIONS AND CAVEATS:
The objectives for this terminated study could not be assessed due to limited data available. (Efficacy parameters were to include BP, heart rate, lipid profile, urine albumin.)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.